CLINICAL TRIAL: NCT04021875
Title: The Effects of Autologous Simple Limbal Epithelial Transplantation.
Brief Title: The Effects of Autologous SLET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904117RINB
Record Dates: First submitted 2019-07-03; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Limbal Stem-cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to prospectively evaluate the therapeutic effects of autologous simple limbal epithelial transplantation for patients with limbal stem cell deficiency. The change of visual acuity, quality of life and so on will be monitored before and after surgery.

DETAILED DESCRIPTION:
Human corneal epithelial cells are stratified squamous cells that cover the corneal surface. These cells are regenerated from cells known as limbal stem cells (LSCs) that grow continuously and proliferate from the limbus. Failure or damage at the limbal zone can occur from hereditary or acquired causes such as ocular burns, trauma, or diseases such as Stevens- Johnson syndrome, leading to limbal stem cell deficiency (LSCD). The treatment of LSCD includes transplantation of healthy limbal tissue or cultured limbal epithelial cells. In the last two decades, cultivated limbal epithelial transplantation (CLET) has been a widely used technique. In 2012, Sangwan and coworkers proposed a novel technique that they named simple limbal epithelial transplantation (SLET) for the treatment of unilateral LSCD1. SLET could have benefits for those centers that do not have the ability to perform cultivated limbal epithelial transplantation (CLET) preparation and could be especially useful for those countries that cannot afford a GMP center. Therefore, SLET is quickly gaining popularity in countries like India. As it is a relatively new technique, its long-term clinical effectiveness (similar to what is observed in CLET) must be noted before determining its actual benefits.Our study aims to prospectively evaluate the therapeutic effects of autologous simple limbal epithelial transplantation for patients with limbal stem cell deficiency. The change of visual acuity, quality of life and so on will be monitored before and after surgery. In this study, the effects of autologous simple limbal epithelial transplantation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-90 years old
2. The lesion eye has at least grade 2 limbal stem cell deficiency
3. The lesion eye has limbal stem cell deficiency causing recurrent corneal erosion and neovascularization ingrowth
4. The symptoms last for at least 6 months and do not improve with medication

Exclusion Criteria:

1. Symptoms improve spontaneously or under medication
2. Someone who can not be examined regularly after the operation
3. Someone with poor prognosis
4. Severe lagophthalmos or trichiasis that has not been corrected
5. Ocular infection

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with limbal stem cell deficiency
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients with clinical success | 6 months
  Clinical success was defined as a completely epithelized, avascular, stable corneal surface. Failure was defined as a recurrence of fibrovascular pannus encroaching on the central cornea, frequent epithelial breakdown or persistent epithelial defects. Kaplan-Meier survival curves were constructed and survival probability calculated using the SPSS software for statistical computing. Focal recurrences of pannus not progressing to the central cornea were not considered as failures and were evaluated separately.

SECONDARY OUTCOMES:
Visual acuity change | 6 months
  Secondary outcome measures included change from baseline visual acuity at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, phD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Republic of China, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Result] Sangwan VS, Basu S, MacNeil S, Balasubramanian D. Simple limbal epithelial transplantation (SLET): a novel surgical technique for the treatment of unilateral limbal stem cell deficiency. Br J Ophthalmol. 2012 Jul;96(7):931-4. doi: 10.1136/bjophthalmol-2011-301164. Epub 2012 Feb 10. PMID 22328817
- [Result] Vazirani J, Ali MH, Sharma N, Gupta N, Mittal V, Atallah M, Amescua G, Chowdhury T, Abdala-Figuerola A, Ramirez-Miranda A, Navas A, Graue-Hernandez EO, Chodosh J. Autologous simple limbal epithelial transplantation for unilateral limbal stem cell deficiency: multicentre results. Br J Ophthalmol. 2016 Oct;100(10):1416-20. doi: 10.1136/bjophthalmol-2015-307348. Epub 2016 Jan 27. PMID 26817481
- [Result] Borroni D, Wowra B, Romano V, Boyadzhieva M, Ponzin D, Ferrari S, Ahmad S, Parekh M. Simple limbal epithelial transplantation: a review on current approach and future directions. Surv Ophthalmol. 2018 Nov-Dec;63(6):869-874. doi: 10.1016/j.survophthal.2018.05.003. Epub 2018 May 22. PMID 29800578